CLINICAL TRIAL: NCT02601508
Title: A Randomized, Parallel Design, Single-center Study to Compare of Surgical Condition and Postoperative Complications With Moderate and Deep Neuromuscular Blockade in Laparoscopic Gastrectomy
Brief Title: Compare of Surgical Condition and Complications With Moderate and Deep NM Block
Acronym: MISPCNUHH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Seongwook Jeong, associate professor, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNUHH-2015-135
Record Dates: First submitted 2015-11-03; First posted 2015-11-10 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Neuromuscular Blockade
Keywords: deep NM block; Surgeon's satisfaction; bridion
MeSH Terms: interventions — Rocuronium; cisatracurium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modarate Blockade Group (Active Comparator): Neuromuscular blocking agent, cis-atracurium will be administered after skin incision and reversal agents, pyridostigmine & glycopyrrolate will be given for the recovery.
  Interventions: Drug: cis-atracurium
- Deep Blockade Group (Experimental): Neuromuscular blocking agent, rocuronium will be administered after skin incision and reversal agent, Sugammadex will be given for the recovery.
  Interventions: Drug: Rocuronium

INTERVENTIONS:
Drug: Rocuronium — Continuous infusion of rocuronium for PTC 1 + Sugammadex
  Other Names: Esmeron®
  Arms: Deep Blockade Group
Drug: cis-atracurium — Intermittent injection of cis-atracurium for TOF 1 + Pyridostigmine & Glycopyrrolate
  Other Names: Nimbex®
  Arms: Modarate Blockade Group

SUMMARY:
This study is designed to evaluate the surgeon's satisfaction with either deep or moderate neuromuscular blockade during laparoscopic gastrectomy surgery and observe the recovery profiles in the recovery room and the ward.The explorative objective of this study is to evaluate the safety profiles of deep and moderate neuromuscular blockades via observation of postoperative complications.

DETAILED DESCRIPTION:
Neuromuscular blocking agents (NMBAs) are frequently using during anesthesia to facilitate tracheal intubation and to improve surgical conditions. In an adequately anesthetized and monitored patient, the presence of one or two responses in the train-of-four (TOF) pattern normally indicates sufficient relaxation for most surgical procedures in general practices. It has been called moderate neuromuscular blockade (mNMB) condition. Nowadays, laparoscopic surgeries have expanded impressively into various areas of surgeries, both in scope and volume. If any hypothetical advantages of deep neuromuscular blockade (dNMB) during laparoscopic surgery turned out to be realized in practice with sufficient supporting evidence, it would become an important anesthetic option for better patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All adult (≥ 20 years of age) patients scheduled for an elective laparoscopic gastrectomy who have signed the written informed consent.

Exclusion Criteria:

* Known allergy to rocuronuim, cisatracurium or sugammadex
* Significant liver or kidney dysfunction
* Any neuromuscular disease
* Pregnant or breast feeding
* Indication for rapid sequence induction
* Inability to give informed consent
* Patients taking any medication with potential interference with neuromuscular transmission

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Surgical rating SCORE(SRS) | every 15 minutes from the pneumoperitoneum, up to 120 minutes till the end of surgery
  excellent (5), good but not optimal (4), moderate (3), poor but acceptable (2) or poor and unacceptable (1)

SECONDARY OUTCOMES:
Respiratory rate | every 15 minutes from the arrival on the recovery room, up to 60 minutes
  Respiratory rate of patient
peripheral arterial oxygen saturation | every 15 minutes from the arrival on the recovery room, up to 60 minutes
  peripheral arterial oxygen saturation(sPO2)
visual analogue scale (VAS) for pain | every 15 minutes from the arrival on the recovery room, up to 60 minutes
  visual analogue scale (VAS) for pain
occurrence of nausea or vomiting | every 15 minutes from the arrival on the recovery room, up to 60 minutes
  occurrence of nausea or vomiting with Rhodes Index
the level of sedation or alertness | every 15 minutes from the arrival on the recovery room, up to 60 minutes
  the level of sedation or alertness with OAA/S scale
Postoperative Quality Recovery Scale (PQRS) | at baseline (the day before surgery), at 1 hour after surgery, at 6 hours after surgery, at 24 hours after surgery and at 7 days after surgery
  physiologic, nociceptive, emotive, cognitive and activities of daily living

CONTACTS AND LOCATIONS:
Overall Officials: SEONGWOOK JEONG, MD, PhD., Principal Investigator — Chonnam University Hospital
Locations (1):
- Chonnam University Hwasun Hospital, Hwasun, South Korea